CLINICAL TRIAL: NCT01942005
Title: EVER/TMC Mutation as Marker of the Risk of Cutaneous Carcinoma in Immunosuppressed Patients,Especially Patients After Organ Transplantation and Patients With HIV Infection
Brief Title: EVER/TMC Mutation as Marker of the Risk of Cutaneous Carcinoma in Immunosuppressed Patients
Acronym: EBVER/TMC
Status: Completed | Type: Observational
Sponsor: Andreas Arnold (Other)
Responsible Party: Sponsor-Investigator, Andreas Arnold, Dr. med. Andreas Arnold, senior physician, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 11/10
Record Dates: First submitted 2013-08-07; First posted 2013-09-13 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Immunosuppression; Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blutsample
Oversight: Data Monitoring Committee: No

SUMMARY:
Detection of mutation / specific polymorphism of the EVER/TMC6 and/or EVER/TMC8 gen.

DETAILED DESCRIPTION:
correlation between possibly detected mutation/specific polymorphism and kind and number of neoplasm, age of patients, UV burden, duration and kind of immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* patients in an immunosuppressive condition either by immunosuppressants or by HIV infection

Exclusion Criteria:

* written informed consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent organ transplatation or patients who have a HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2010-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Detection of mutation / specific polymorphism of the EVER/TMC6 and/or EVER/TMC8 gen. | 7 years

SECONDARY OUTCOMES:
correlation between possibly detected mutation/specific polymorphism of the EVER/TMC6 and/or EVER/TMC8 gen and a composite of kind and number of neoplasm, age of patients, UV burden, duration and kind of immunosuppression. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Arnold, MD, Principal Investigator — University Hospital Basel, Dermatology, CH-4031 Basel
Locations (1):
- University Hospital Basel, Dermatology, Basel, Canton of Basel-City, Switzerland